CLINICAL TRIAL: NCT07336745
Title: Recovery Effects of Electrical Muscle Stimulation After Climbing-Induced Fatigue: A Randomized Crossover Trial
Brief Title: EMS Recovery Effects in Sport Climbing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TSA-2019-4786
Record Dates: First submitted 2025-12-17; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2020-11

CONDITIONS: Exercise-Induced Fatigue; Forearm Muscle Fatigue
Keywords: Sport climbing; Forearm fatigue; Electrical muscle stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMS Recovery (EMSr) Arm (Experimental): Participants completed a standardized climbing fatigue protocol consisting of 15 sets of 1-minute climbs followed by 1-minute rest on a TensionBoard route (IRCRA grade 15). Immediately after the fatigue protocol, participants underwent Electrical Muscle Stimulation-based Recovery (EMSr). EMS was applied to the forearm flexor muscles (flexor carpi radialis, palmaris longus, flexor carpi ulnaris) using a Chattanooga Wireless Professional 4CH device with 5×5 cm electrodes. The "Active Recovery" program (2-4-6-5-4-3-2-1 Hz; 50 minutes) was used. Stimulation intensity was individually adjusted to elicit visible muscle contraction without discomfort.The EMSr intervention was designed to facilitate local muscle recovery, maintain climbing-specific performance (total move count, isometric hang time), and reduce performance decrements compared to passive rest.
  Interventions: Device: Electrical Muscle Stimulation
- Passive Recovery (PASr) Arm (No Intervention): Participants completed the same standardized climbing fatigue protocol (15 × 1-minute climbs with 1-minute rest on a TensionBoard route, IRCRA grade 15). Immediately after the fatigue protocol, participants underwent passive recovery (PASr), consisting of 50 minutes of seated rest. No active muscle stimulation or exercise was performed during this period.
  The PASr arm serves as a control condition to evaluate the effects of EMS-based recovery on climbing-specific performance metrics.

INTERVENTIONS:
Device: Electrical Muscle Stimulation — This intervention specifically targets the forearm flexor muscles (flexor carpi radialis, palmaris longus, flexor carpi ulnaris) using low-frequency electrical stimulation to promote local muscle recovery after climbing-induced fatigue. The protocol uses a 50-minute "Active Recovery" program (2-4-6-5-4-3-2-1 Hz) applied via a device, with intensity individually adjusted to elicit visible muscle contraction without discomfort. Unlike general active recovery or passive rest, this intervention provides localized neuromuscular stimulation designed to preserve climbing-specific performance metrics such as total move count and weighted isometric hang time.
  Arms: EMS Recovery (EMSr) Arm

SUMMARY:
Sport climbing often requires athletes to perform repeated climbing efforts with short rest periods. Over time, fatigue can build up in the muscles of the arms and forearms, which may reduce performance and increase the difficulty of continuing to climb at the same level.

This study aims to better understand different recovery methods that climbers may use between climbing efforts. Specifically, the study compares two recovery approaches: electrical muscle stimulation-based recovery and passive recovery (resting while seated).

In this study, adult male sport climbers will complete a structured climbing task designed to induce fatigue. After the climbing task, participants will receive one of the two recovery methods. On a separate study visit, they will complete the same procedure using the other recovery method. The order of the recovery methods will be randomized, and there will be a break of one week between sessions.

During the study sessions, researchers will record climbing-related performance measures, simple strength and endurance tasks, heart rate, and how hard the participants feel they are working. The information collected will help researchers better understand recovery strategies used in climbing and may inform training and recovery practices for athletes in the future.

Participation in the study is voluntary, and all procedures are conducted under controlled laboratory conditions.

DETAILED DESCRIPTION:
Sport climbing places high and repetitive demands on the forearm muscles, which are required to sustain repeated gripping and pulling actions with limited recovery time. During prolonged or repeated climbing bouts, local muscular fatigue can accumulate, potentially affecting endurance and movement quality. Competitive climbers are particularly exposed to these demands, as competitions often involve multiple rounds performed within the same day with short rest intervals. For this reason, recovery strategies that can be applied between climbing efforts are of practical relevance in both training and competition settings.

Electrical muscle stimulation (EMS) is a recovery modality that delivers low-intensity electrical impulses to skeletal muscle, producing rhythmic, involuntary contractions. EMS has been used in various sport and rehabilitation contexts as a low-effort method that can be applied without additional mechanical load. However, its application as an inter-bout recovery strategy in sport climbing has not been sufficiently characterized under controlled, climbing-specific conditions.

This study is designed as a randomized crossover trial to compare EMS-based recovery (EMSr) and passive recovery (PASr) following a standardized climbing fatigue protocol. Advanced male sport climbers will participate in two experimental sessions separated by a one-week washout period. In each session, participants will complete the same climbing fatigue protocol, followed by one of the two recovery conditions, with the order of recovery methods randomized.

The fatigue protocol consists of repeated climbing bouts performed on a standardized training wall using a fixed route of defined difficulty. This protocol is intended to elicit localized forearm fatigue under reproducible conditions. Following completion of the fatigue protocol, participants will undergo either EMS applied to the forearm muscles for a fixed duration or passive recovery involving seated rest without additional intervention.

Climbing-related performance measures, muscular endurance tasks, cardiovascular responses, and ratings of perceived exertion will be recorded at predefined time points before and after the recovery period. These measurements are included to characterize physiological and performance-related responses associated with each recovery condition.

The crossover design allows each participant to serve as their own control, thereby reducing inter-individual variability and enabling a direct comparison of recovery approaches under standardized conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male climbers aged 30-36 years.
* At least 3 years of continuous climbing experience, training 3-4 times per week.
* Ability to climb at least IRCRA grade 15 (French 6a) routes.
* In good general health and able to safely perform high-intensity climbing.
* Willing to provide written informed consent and follow study instructions.

Exclusion Criteria:

* Participation in other sports with high training loads that could interfere with the study.
* Any injury, medical condition, or musculoskeletal problem that limits climbing performance.
* Use of medications or supplements that could affect muscle performance or recovery.
* Inability to comply with study procedures, including the climbing and recovery protocols.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Total Move Count During the TensionBoard Fatigue Test Following Recovery Intervention | Immediately after the 50-minute recovery period following the fatigue protocol.
  Total move count represents the number of hand movements completed by each participant during the TensionBoard Fatigue Test, which consists of 15 sets of 1-minute climbs with 1-minute rests on a standardized route (IRCRA grade 15). This measure assesses climbing-specific performance and endurance, reflecting the ability to sustain high-intensity climbing efforts after the fatigue protocol. Move count is recorded for each set, and the change from baseline (pre-recovery) to post-recovery is used to evaluate the effectiveness of the intervention (EMS recovery vs. passive rest).

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Faculty of Sport Sciences, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from this study, including climbing performance metrics, recovery protocol details, and anthropometric measurements, will be made available to other researchers upon reasonable request. Requests should be submitted to the corresponding author (Tuba Melekoğlu, tmelekoglu@akdeniz.edu.tr) and will require a data use agreement outlining the purpose of analysis, protection of participant confidentiality, and acknowledgment of the original study. Data will be available for academic and non-commercial research purposes for 5 years following publication of the study results.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start Date: Upon publication of the study results (estimated June 2026) End Date: 5 years after publication (estimated June 2031)
Access Criteria: Who can access: Qualified researchers from academic or non-commercial research institutions who submit a reasonable request and agree to a data use agreement.
  What they can access: De-identified individual participant data, including climbing performance metrics (total move count, isometric hang time, push-up and sit-up performance), anthropometric measurements, and details of the recovery protocols (EMS and passive recovery). Supporting documentation, such as the study protocol and data dictionaries, will also be provided.
  How they can access: Requests must be submitted to the corresponding author (Tuba Melekoğlu, tmelekoglu@akdeniz.edu.tr). Upon approval and signing of a data use agreement, datasets and supporting information will be shared electronically in a secure format.